CLINICAL TRIAL: NCT01041183
Title: The Effect of Oral and Intravenous Ramosetron During Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nasea-LC
Record Dates: First submitted 2009-12-30; First posted 2009-12-31 (Estimated); Last update posted 2009-12-31 (Estimated); Status verified 2009-11

CONDITIONS: Nausea; Vomiting; Laparoscopic Cholecystectomy
Keywords: Oral plus IV ramosetron may be more effective than; IV ramosetron and oral ramosetron for the prophylaxis of; PONV after laparoscopic cholecystectomy
MeSH Terms: conditions — Nausea; Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- group I (Active Comparator): 0.3 mg IV ramosetron
  Interventions: Drug: intravenous ramosetron
- group II (Active Comparator): 0.1 mg oral ramosetron
  Interventions: Drug: oral ramosetron
- group III (Active Comparator): 0.1 mg oral ramosetron plus 0.3 mg IV ramosetron
  Interventions: Drug: oral and IV ramosetron

INTERVENTIONS:
Drug: intravenous ramosetron — 0.3 mg IV ramosetron (group I)
  Arms: group I
Drug: oral ramosetron — 0.1 mg oral ramosetron (group II)
  Arms: group II
Drug: oral and IV ramosetron — 0.1 mg oral ramosetron plus 0.3 mg IV ramosetron (group III).
  Arms: group III

SUMMARY:
Patients undergoing general anesthesia for laparoscopic cholecystectomy have a high risk of postoperative nausea and vomiting (PONV). The investigators investigated the effect of oral and IV ramosetron on PONV prophylaxis after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients, 25-65 years, electivelaparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* GI disease, pregnant or menstruating, history of motion sickness and/or postoperative emesis, antiemetics within 24 h before surgery

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV | postoperative 0-48 h

CONTACTS AND LOCATIONS:
Locations (1):
- Jung-Hee Ryu, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Ryu JH, Jeon YT, Hwang JW, Oh AY, Moon JY, Ro YJ, Kim CS, Chen C, Apfel CC, Do SH. Intravenous, oral, and the combination of intravenous and oral ramosetron for the prevention of nausea and vomiting after laparoscopic cholecystectomy: a randomized, double-blind, controlled trial. Clin Ther. 2011 Sep;33(9):1162-72. doi: 10.1016/j.clinthera.2011.07.018. PMID 21856001